CLINICAL TRIAL: NCT04387747
Title: Evaluation Of Sarcopenia In Stroke Patients
Brief Title: Evaluation of Sarcopenia in Patients With Stroke
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Aydın, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: ıstPMRTRH-SRCPN
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-05

CONDITIONS: Sarcopenia; Stroke
Keywords: sarcopenia; stroke
MeSH Terms: conditions — Sarcopenia; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SARCOPENIA IN STROKE PATIENTS — Demographic characteristics, duration of stroke, sarcopenia presence,thigh circumference , Hand grip strength , TANITA BIA analysis

SUMMARY:
The aim of this study is to investigate the prevalence of sarcopenia in stroke patients; to determine the relationship between sarcopenia and duration of stroke, age, gender, etiology of stroke, ambulation status, spasticity, nutrition and malnutrition

DETAILED DESCRIPTION:
Sarcopenia was defined as a loss of skeletal muscle mass and decreased muscle strength. The purpose of this study was to investigate the prevalence of sarcopenia following stroke, to investigate the relationship between sarcopenia and duration of stroke, age, sex, etiology of stroke, ambulation status, spasticity, nutrition and malnutrition. Demographic characteristics, duration of stroke, sarcopenia presence (walking speed ≥ 0.8 m / s, SARC-F score ≥4, short physical performance battery score ≤ 8, thigh circumference <33cm (The data for Turkey) <31cm (European data)) were recorded. Hand grip strength (jamar) measured from the intact hand and TANITA BIA analysis were planned for all patients.

Ambulation level with Functional Ambulation Classification (FAC), nutritional status with 24-hour dietary recall (24HR) method, diagnosis of malnutrition with Glim Criteria, spasticity with Modified Ashworth Scale, motor development for stroke patient Brunnstrom staging, screening for frailty with Frail questionnaire activity of daily living were evaluated with Barthel Index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stroke (Stroke duration > 3 months)
* Patients with a FAC score > 3

Exclusion Criteria:

* Patients unable to cooperate
* Other diseases that cause gait disorders such as neuromuscular disease, cardiopulmonary problems.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient stroke cases
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Classification (FAC) | 1 interview day
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. FAC stage 0 indicates the non-functional ambulation, and stage 5 indicates the independent walking at each speed and on ground.
24-hour dietary recall (24HR) method | 1 interview day
  24-hour dietary recall method consists of precisely recalling, describing and quantifying the intake of foods and beverages consumed during the day before the interview, from the first intake in the morning until the last foods or beverages consumed at night.
Glim Criteria | 1 interview day
  The five criteria for malnutrition include non-volitional weight loss, low body mass index, and reduced muscle mass as phenotypic criteria, and reduced food intake/assimilation and inflammation/disease burden as etiologic criteria. It is proposed that the diagnosis of malnutrition be based upon the presence of at least one phenotypic criterion and one etiologic criterion.
sarcopenia | 1 interview day
  The walking speed ≥0.8 m / s, SARC-F score ≥4, short physical performance battery score ≤ 8, thigh circumference <33cm.
EQ-5D | 1 interview day
  EQ-5D-3L is used to evaluate the quality of life. This scale scores five health conditions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) through evaluation in 3 levels (no problems, some problems, extreme problems).

SECONDARY OUTCOMES:
Barthel index | 1 interview day
  The Barthel Index measures the activity limitations in patients with neuromuscular disease. The Barthel Index are assessed, including toileting, bathing, eating, dressing, continence, transfers, and ambulation. A client scoring 0 points would be dependent in all assessed activities of daily living, whereas a score of 100 would reflect independence in these activities.
Brunnstrom's staging | 1 interview day
  Brunnstrom's staging is used to evaluate the sequence of motor development and reorganization of the brain after stroke in six stages. Stage 1: Flaccidity; Stage 2: Spasticity Appears; Stage 3: Increased Spasticity; Stage 4: Decreased Spasticity; Stage 5: Spasticity Continues to Decrease; Stage 6: Spasticity Disappears and Coordination Reappears.
Modified Ashworth Scale | 1 interview day
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Scoring: 0: No increase in muscle tone; 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2: More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved; 3: Considerable increase in muscle tone, passive movement difficult; 4: Affected part(s) rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scherbakov N, Sandek A, Doehner W. Stroke-related sarcopenia: specific characteristics. J Am Med Dir Assoc. 2015 Apr;16(4):272-6. doi: 10.1016/j.jamda.2014.12.007. Epub 2015 Feb 10. PMID 25676847
- [Background] Ryan AS, Ivey FM, Serra MC, Hartstein J, Hafer-Macko CE. Sarcopenia and Physical Function in Middle-Aged and Older Stroke Survivors. Arch Phys Med Rehabil. 2017 Mar;98(3):495-499. doi: 10.1016/j.apmr.2016.07.015. Epub 2016 Aug 13. PMID 27530769
- [Derived] Aydin T, Kesiktas FN, Oren MM, Erdogan T, Ahisha YC, Kizilkurt T, Corum M, Karacan I, Ozturk S, Bahat G. Sarcopenia in patients following stroke: an overlooked problem. Int J Rehabil Res. 2021 Sep 1;44(3):269-275. doi: 10.1097/MRR.0000000000000487. PMID 34356039